CLINICAL TRIAL: NCT01259115
Title: A Single Center, Randomized, Double-Blind, Crossover Study to Assess Buprenorphine Accumulation and Description of Its Metabolites During Co-Medication of BTDS and Ketoconazole, Used As a CYP3A4 Inhibitor, in Healthy Subjects
Brief Title: Buprenorphine Accumulation and Description of Its Metabolites During Co-Medication of Buprenorphine Transdermal System (BTDS) and Ketoconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: BUP1009
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Healthy subjects; Opioid; Transdermal
MeSH Terms: interventions — Buprenorphine; Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): BTDS 10 with ketoconazole 200 mg tablets twice daily in period 1 and BTDS 10 with ketoconazole placebo tablets twice daily in period 2.
  Interventions: Drug: Buprenorphine transdermal patch; Drug: Ketoconazole tablet; Drug: Placebo to match ketoconazole tablet
- Sequence B (Experimental): BTDS 10 with ketoconazole placebo tablets twice daily in period 1 and BTDS 10 with ketoconazole 200 mg twice daily in period 2.
  Interventions: Drug: Buprenorphine transdermal patch; Drug: Ketoconazole tablet; Drug: Placebo to match ketoconazole tablet

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine 10 mcg/hour patch applied transdermally for 7-day wear.
  Other Names: Butrans™
Drug: Ketoconazole tablet — Ketoconazole 200 mg tablets taken orally twice daily.
Drug: Placebo to match ketoconazole tablet — Placebo to match ketoconazole 200 mg tablets taken orally twice daily.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of buprenorphine and its metabolites in the presence and absence of ketoconazole.

DETAILED DESCRIPTION:
To assess the pharmacokinetics of buprenorphine and its metabolites (nor-buprenorphine, buprenorphine 3 glucuronide and nor-buprenorphine glucuronide) in the presence and absence of ketoconazole.

Safety evaluation of BTDS and ketoconazole in healthy subjects.

ELIGIBILITY:
Inclusion Criteria Include:

* Males and females aged 18 to 54 years.
* Demonstrate CYP 3A4 inhibition by ketoconazole with the erythromycin breath test (EBT) probe during the screening period.
* Female subjects who are surgically sterile or at least two years postmenopausal.
* Have a body weight ranging from 60 to 100 kilograms (kg), and are within 15% of optimum for height and body frame, as determined from parameters of the Metropolitan Life Index.
* Agree not to use any medication, including over-the-counter (OTC) medications, vitamins, mineral or herbal supplements, during the course of the study and for at least 7 days prior to the start of the study.
* Generally in good health as evidenced by lack of significant abnormal finding(s) in medical history, physical examination, clinical laboratory tests, vital signs, and electrocardiogram (ECG).
* Willing to follow dietary restrictions, including abstention from grapefruit, herbal dietary supplements especially those containing St. John's Wort, and caffeine containing products.
* Willing to refrain from strenuous exercise or contact sports during the study

Exclusion Criteria Include:

* Any history of hypersensitivity to buprenorphine, any excipient of BTDS, ketoconazole, or other opioids, psychotropic or hypnotic drugs.
* Any medical or surgical conditions that might interfere with transdermal drug absorption (eg skin lesions at site of application), gastrointestinal drug absorption (eg, delayed gastric emptying, malabsorption syndromes), distribution (eg, obesity), metabolism, or excretion (eg, hepatitis, glomerulonephritis).
* Any history of significant active medical illness such as:
* History or presence of liver disease or injury as indicated by increase of aspartate transaminase (AST) or alanine transaminase (ALT) or bilirubin above the normal levels
* History or presence of renal insufficiency as indicated by abnormal creatinine or blood urea nitrogen (BUN) or abnormal urinary constituent (eg, albumin).
* Any other clinically significant laboratory abnormalities.
* At risk of transmitting infection via blood samples such as:
* producing a positive human immunodeficiency virus (HIV) test at screening or having participated in a high risk activity for contracting HIV
* producing a positive Hepatitis B surface antigen test at screening
* producing a positive Hepatitis C antibody test at screening.
* Any personal or family history of prolonged QT interval or disorders of cardiac rhythm, including heartbeat below 45, unless agreed upon by sponsor.
* Females who are breastfeeding.
* Females with a positive serum or urine pregnancy test at screening or prior to dosing, respectively.

Other protocol-specific exclusion/inclusion criteria may apply.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2002-10; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, New Orleans, Louisiana, United States

REFERENCES:
- [Result] Kapil RP, Cipriano A, Michels GH, Perrino P, O'Keefe SA, Shet MS, Colucci SV, Noveck RJ, Harris SC. Effect of ketoconazole on the pharmacokinetic profile of buprenorphine following administration of a once-weekly buprenorphine transdermal system. Clin Drug Investig. 2012 Sep 1;32(9):583-92. doi: 10.1007/BF03261913. PMID 22845044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21-Oct-2002 (first subject, first visit) to 20-Jun-2003 (last subject, last visit). Study conducted at 1 site in New Orleans, LA.
Pre-assignment Details: Healthy male and female subjects aged 18 to 54 years, demonstrating successful inhibition of CYP3A4 using the EBT (erythromycin breath test) probe were randomized.
Groups:
- Sequence A: BTDS 10 With Ketoconazole (Test) First: Period 1: Buprenorphine transdermal system (BTDS) 10 with ketoconazole 200 mg tablets twice daily (Test) first;
  Washout Period of 4 to 18 days;
  Period 2: BTDS 10 with ketoconazole placebo tablets twice daily.
- Sequence B: BTDS 10 With Placebo (Reference) First: Period 1: Buprenorphine transdermal system (BTDS) 10 with ketoconazole placebo tablets twice daily (Reference) first
  Washout Period of 4 to 18 days;
  Period 2: BTDS 10 with ketoconazole 200 mg tablets twice daily.
Period: Period 1
Arm/Group | Sequence A: BTDS 10 With Ketoconazole (Test) First | Sequence B: BTDS 10 With Placebo (Reference) First
Started | 10 | 10
Completed | 7 | 9
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Period: Washout Period of 4 to 18 Days
Arm/Group | Sequence A: BTDS 10 With Ketoconazole (Test) First | Sequence B: BTDS 10 With Placebo (Reference) First
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence A: BTDS 10 With Ketoconazole (Test) First | Sequence B: BTDS 10 With Placebo (Reference) First
Started | 7 | 9
Completed | 6 | 9
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects received BTDS 10 with ketoconazole 200 mg or ketoconazole placebo tablets twice daily in period 1; Washout Period for 4 to 18 days; Subjects received BTDS 10 with ketoconazole 200 mg or ketoconazole placebo tablets twice daily in period 2.
Arm/Group | Overall Study
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: AUCt of Buprenorphine With and Without Ketoconazole.
Description: AUCt (area under the plasma concentration-time curve from hour 0 to the last measurable plasma concentration) of buprenorphine transdermal patch 10 with and without ketoconazole 200 mg oral twice daily.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or Ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: The full analysis population for pharmacokinetics was defined as those subjects who received at least 1 dose of study drug and did not have any incidents of emesis for at least 12 hours from dosing during at least 1 period and had at least 1 valid pharmacokinetic metric.
Measure: Mean (Standard Deviation); unit: pg/mL*h
Groups:
- BTDS 10 With Ketoconazole: Period 1: BTDS 10 with ketoconazole 200 mg tablets twice daily; Washout: Day 12 to 15; Period 2: BTDS 10 with ketoconazole placebo tablets twice daily.
- BTDS 10 With Ketoconazole Placebo: Period 1: BTDS 10 with ketoconazole placebo tablets twice daily; Washout: Day 12 to 15; Period 2: BTDS 10 with ketoconazole 200 mg twice daily.
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 18 | 16
pg/mL*h | 16354.8 (6197.3) | 16627.9 (5559.7)

2. Primary Outcome: AUCinf of Buprenorphine With and Without Ketoconazole.
Description: AUCinf (the area under the plasma-concentration time course profile from time 0 [dosing] to infinity) of buprenorphine transdermal patch 10 with and without ketoconazole 200 mg oral twice daily.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg /mL•h
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 13 | 9
pg /mL•h | 18238.5 (6624.5) | 19012.5 (6599.2)

3. Primary Outcome: Cmax of Buprenorphine With and Without Ketoconazole.
Description: Cmax (maximum observed plasma concentration) of buprenorphine transdermal patch 10 with and without ketoconazole 200 mg oral tablets twice daily,
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: The full analysis population for pharmacokinetics was defined as those subjects who received at least 1 dose of study drug and did not have any incidents of emesis for at least 12 hours from dosing during at least 1 period and had at least 1 valid PK metric.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 18 | 16
pg/mL | 142.2 (53.7) | 145.5 (48.7)

4. Primary Outcome: AUCt of Nor-buprenorphine With and Without Ketoconazole
Description: For nor-buprenorphine pharmacokinetic metric, AUCt (area under the plasma concentration-time curve from hour 0 to the last measurable plasma concentration).
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL*h
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 16 | 11
pg/mL*h | 5091.0 (3208.3) | 3207.8 (1746.4)

5. Secondary Outcome: CYP3A4 Inhibition by Observation of Plasma Nor-buprenorphine Production Assessed by the Erythromycin Breath Test.
Description: As part of subject screening, Erythromycin Breath Tests (EBT) were done on all potential subjects (enrolled population). CYP 3A4 inhibition was calculated by taking the difference of the baseline 14C erythromycin metabolism, subtracting the 14C erythromycin metabolism during ketoconazole treatment, dividing this difference by the baseline 14C erythromycin metabolism, and multiplying by 100 to express results in the form of percent inhibition. CYP3A4 inhibition was only done when subjects were on ketoconazole.
Time Frame: One time at screening and one time during ketoconazole treatment
Population: Enrolled Population: All subjects who participated in the study. CYP3A4 Inhibition was only done when subjects were on Ketoconazole.
Measure: Mean (Standard Deviation); unit: Percentage of participants
Groups:
- All Subjects: Subjects who received BTDS with Ketoconazole treatment
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Percentage of participants
  All subjects [N = 20] | 64.49 (15.69)
  Inhibition ≤ 50% [n = 4] | 37.50 (4.11)
  Inhibition >50% but ≤ 70% [n = 8] | 64.50 (4.61)
  Inhibition > 70% [n = 8] | 77.98 (3.94)

6. Primary Outcome: AUCinf of Nor-buprenorphine With and Without Ketoconazole
Description: For nor-buprenorphine pharmacokinetic metric, AUCinf (the area under the plasma-concentration time course profile from time 0 [dosing] to infinity).
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL*h
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 1 | 0
pg/mL*h | 6767.9 (0) |

7. Primary Outcome: Cmax of Nor-buprenorphine With and Without Ketoconazole
Description: For nor-buprenorphine pharmacokinetic metric, Cmax (maximum observed plasma concentration), log transformed data were analyzed.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 16 | 11
pg/mL | 63.4 (25.9) | 44.6 (11.1)

8. Primary Outcome: AUCt of Nor-buprenorphine Glucuronide With and Without Ketoconazole
Description: For nor-buprenorphine glucuronide pharmacokinetic metrics, AUCt (area under the plasma concentration-time curve from hour 0 to the last measurable plasma concentration), log transformed data were analyzed.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL*h
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 18 | 16
pg/mL*h | 21376.9 (9808.2) | 15840.5 (5034.5)

9. Primary Outcome: AUCinf of Nor-buprenorphine Glucuronide With and Without Ketoconazole
Description: For nor-buprenorphine glucuronide pharmacokinetic metrics, AUCinf (the area under the plasma-concentration time course profile from time 0 [dosing] to infinity) log transformed data were analyzed.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL*h
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 0 | 3
pg/mL*h |  | 17318.9 (657.2)

10. Primary Outcome: Cmax of Nor-buprenorphine Glucuronide With and Without Ketoconazole
Description: For nor-buprenorphine glucuronide pharmacokinetic metric, Cmax (maximum observed plasma concentration), log transformed data were analyzed.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 18 | 16
pg/mL | 218.2 (99.4) | 141.9 (47.6)

11. Primary Outcome: AUCt of Buprenorphine-3-glucuronide With and Without Ketoconazole
Description: For buprenorphine-3-glucuronide pharmacokinetic metric, AUCt (area under the plasma concentration-time curve from hour 0 to the last measurable plasma concentration), log transformed data were analyzed.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL*h
Groups:
- BTDS 10 With Ketoconazole: BTDS 10 with ketoconazole 200 mg tablets twice daily
- BTDS 10 With Ketoconazole Placebo: Buprenorphine-3-glucuronide was not measured in the plasma during treatment
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 5 | 0
pg/mL*h | 342.4 (488.2) |

12. Primary Outcome: AUCinf of Buprenorphine-3-glucuronide With and Without Ketoconazole
Description: For buprenorphine-3-glucuronide pharmacokinetic metric, AUCinf (the area under the plasma-concentration time course profile from time 0 [dosing] to infinity), log transformed data were analyzed.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Cmax of Buprenorphine-3-glucuronide With and Without Ketoconazole
Description: For buprenorphine-3-glucuronide pharmacokinetic metric, Cmax (maximum observed plasma concentration), log transformed data were analyzed.
  Period 1, subjects wore BTDS 10 patch between days 3 and 10 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 1 and 11. Washout period of 4 to 18 days. Period 2, subjects wore BTDS 10 patch between days 19 and 26 and took ketoconazole (200 mg orally twice daily) or ketoconazole placebo (orally twice daily) between days 17 and 27.
Time Frame: BTDS Days 3, 10, 19, and 26; ketoconazole or placebo Days 9 and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 5 | 0
pg/mL | 88.5 (85.6) |

14. Secondary Outcome: The Number of Participants With Adverse Events (AEs) as a Measure of Safety.
Description: Safety assessments consisted of monitoring and recording medical history, physical examinations, vital signs (including temperature, heart rate, blood pressure and respiratory rate), reports of adverse experiences, and laboratory abnormalities (including electrocardiogram [ECG]).
Time Frame: The first day of study drug administration to 30 days after the last dose of study drug.
Population: Safety Population: Safety analyses were performed on all subjects who received at least 1 dose of study drug and for whom at least 1 postdose safety observation was recorded.
Measure: Number; unit: participants
Groups:
- BTDS 10 With Ketoconazole: Buprenorphine transdermal system (BTDS) 10 with ketoconazole 200 mg tablets twice daily.
- BTDS 10 With Ketoconazole Placebo: Buprenorphine transdermal system (BTDS) 10 with ketoconazole placebo oral tablets twice daily.
Arm/Group | BTDS 10 With Ketoconazole | BTDS 10 With Ketoconazole Placebo
Number analyzed (Participants) | 19 | 17
participants
  Deaths | 0 | 0
  Serious Adverse Events | 0 | 0
  Adverse Events in 4% or more of subjects | 19 | 16

ADVERSE EVENTS:
Time Frame: All adverse events during the course of the study were collected and were to be followed until resolution or for 30 days after the last dose of study drug. Serious adverse events were followed until the event resolved or sequelae stabilized.
Description: AEs were learned of by spontaneous reports, subject interview, and daily diary
Groups:
- BTDS With Ketoconazole: Subjects who were treated with buprenorphine transdermal patch 10 mcg/hour with ketoconazole 200 mg oral tablets twice daily.
- BTDS With Placebo: Subjects who were treated with buprenorphine transdermal patch 10 mcg/hour with ketoconazole placebo oral tablets twice daily.
Arm/Group | BTDS With Ketoconazole | BTDS With Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 19/19 | 16/17
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BTDS With Ketoconazole (N=19) | BTDS With Placebo (N=17)
Cardiospasm (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Abdominal pain (General disorders) | 1 | 1
Back pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Headache (General disorders) | 5 | 3
Ecchymosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Creatinine increased (Metabolism and nutrition disorders) | 2 | 0
Infection (Infections and infestations) | 1 | 0
Accidental Injury (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 6 | 5
Somnolence (Nervous system disorders) | 0 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema at site (Skin and subcutaneous tissue disorders) | 13 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus at site (Skin and subcutaneous tissue disorders) | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Dry eyes (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Urination impaired (Renal and urinary disorders) | 1 | 1
Leukorrhea (Renal and urinary disorders) | 1 | 0
Vasodilatation (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days